CLINICAL TRIAL: NCT06771622
Title: Phase Ib/IIa, Open-label, Multicenter, Dose Escalation, and Dose Expansion Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Antitumor Activity of HCB101 in Combination With Multiple Agents in Subjects With Advanced Solid Tumors
Brief Title: Safety and Efficacy of HCB101 in Combination With Multiple Agents in Patients With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: FBD Biologics Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCB101-201
Record Dates: First submitted 2025-01-08; First posted 2025-01-13 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-04

CONDITIONS: Solid Cancer
MeSH Terms: interventions — Trastuzumab; pertuzumab; Oxaliplatin; Capecitabine; Ramucirumab; Paclitaxel; Bevacizumab; Cetuximab; Irinotecan; Leucovorin; Fluorouracil; toripalimab; Albumin-Bound Paclitaxel; pembrolizumab; Carboplatin; Etoposide; atezolizumab; trastuzumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (14):
- Cohort 1: HCB101+Trastuzumab+Pertuzumab+CAPEOX (Experimental): HCB101: QW Trastuzumab: 8 mg/kg IV loading dose on Day 1 of cycle 1, then 6 mg/kg IV every 21 days; Pertuzumab: 840 mg IV on Day 1, cycled every 21 days; Oxaliplatin: 130 mg/m2 IV on Day 1, cycled every 21 days; Capecitabine: 1000 mg/m2 PO BID on Days 1-14, cycled every 21 days;
  Interventions: Drug: HCB101; Drug: Trastuzumab; Drug: Pertuzumab; Drug: Oxaliplatin; Drug: Capecitabine
- Cohort 2: HCB101+Ramucirumab+Paclitaxel (Experimental): HCB101: QW Ramucirumab: 8 mg/kg IV on Days 1 and 15, cycled every 28 days; Paclitaxel: 80 mg/m2 IV on Days 1, 8, and 15, cycled every 28 days;
  Interventions: Drug: HCB101; Drug: Ramucirumab; Drug: Paclitaxel
- Cohort 3a: HCB101 + Bevacizumab + FOLFIRI/ mFOLFOX6 (Experimental): HCB101: QW Bevacizumab 5 mg/kg IV on D1, Q2W
  FOLFIRI:
  Irinotecan 180 mg/m2 IV on D1, Q2W Leucovorin 400 mg/m2 IV on D1, Q2W 5-FU 400 mg/m2 IV on D1, then 1200 mg/m2/day on D2 and D3 (total 2400 mg/m2), Q2W
  mFOLFOX6: Oxaliplatin 85 mg/m2 IV on D1, Q2W Leucovorin 400 mg/m2 IV on D1, Q2W 5-FU 400 mg/m2 IV on D1, then 1200 mg/m2/day on D2 and D3 (total 2400 mg/m2), Q2W
  Interventions: Drug: HCB101; Drug: Oxaliplatin; Drug: Bevacizumab; Drug: Irinotecan; Drug: Leucovorin; Drug: 5-FU; Drug: Pembrolizumab
- Cohort 3b: HCB101 + Cetuximab + FOLFIRI/ mFOLFOX6 (Experimental): HCB101: QW Cetuximab 400 mg/m2 IV on D1, then 250 mg/m2, weekly
  FOLFIRI:
  Irinotecan 180 mg/m2 IV on D1, Q2W Leucovorin 400 mg/m2 IV on D1, Q2W 5-FU 400 mg/m2 IV on D1, then 1200 mg/m2/day on D2 and D3 (total 2400 mg/m2), Q2W
  mFOLFOX6: Oxaliplatin 85 mg/m2 IV on D1, Q2W Leucovorin 400 mg/m2 IV on D1, Q2W 5-FU 400 mg/m2 IV on D1, then 1200 mg/m2/day on D2 and D3 (total 2400 mg/m2), Q2W
  Interventions: Drug: HCB101; Drug: Oxaliplatin; Drug: Cetuximab; Drug: Irinotecan; Drug: Leucovorin; Drug: 5-FU
- Cohort 3c: HCB101 + Ramucirumab + FOLFIRI (Experimental): HCB101: QW Ramucirumab 8 mg/kg IV on D1 and 15, Q4W
  FOLFIRI:
  Irinotecan 180 mg/m2 IV on D1, Q2W Leucovorin 400 mg/m2 IV on D1, Q2W 5-FU 400 mg/m2 IV on D1, then 1200 mg/m2/day on D2 and D3 (total 2400 mg/m2), Q2W
  Interventions: Drug: HCB101; Drug: Ramucirumab; Drug: Irinotecan; Drug: Leucovorin; Drug: 5-FU
- Cohort 3d: HCB101 + mFOLFOX6 (Experimental): HCB101: QW
  mFOLFOX6: Oxaliplatin 85 mg/m2 IV on D1, Q2W Leucovorin 400 mg/m2 IV on D1, Q2W 5-FU 400 mg/m2 IV on D1, then 1200 mg/m2/day on D2 and D3 (total 2400 mg/m2), Q2W
  Interventions: Drug: HCB101; Drug: Oxaliplatin; Drug: Leucovorin; Drug: 5-FU
- Cohort 4: HCB101 + Pembrolizumab/Toripalimab + albumin-bound paclitaxel (Experimental): HCB101, QW Pembrolizumab 200 mg IV on D1, Q3W or Toripalimab 240 mg IV on D1, Q3W Albumin-bound paclitaxel 100 mg/m2 on D1, 8, 15, Q4W or 125 mg/m2 IV on D1, D8, Q3W
  Interventions: Drug: HCB101; Drug: Toripalimab; Drug: Albumin-bound paclitaxel; Drug: Pembrolizumab
- Cohort 5: HCB101 + Pembrolizumab + CAPEOX (Experimental): HCB101, QW Pembrolizumab 200 mg IV on D1, Q3W Oxaliplatin 130 mg/m2 IV on D1, Q3W Capecitabine 1000 mg/m2 PO BID on D1-14, Q3W
  Interventions: Drug: HCB101; Drug: Oxaliplatin; Drug: Capecitabine; Drug: Pembrolizumab
- Cohort 6a: HCB101 + Pembrolizumab (Experimental): HCB101, QW Pembrolizumab 200 mg IV on D1, Q3W
  Interventions: Drug: HCB101; Drug: Pembrolizumab
- Cohort 6b: HCB101 + Pembrolizumab + Cetuximab (Experimental): HCB101, QW Pembrolizumab 200 mg IV on D1, Q3W Cetuximab 400 mg/m2 IV on D1, then 250 mg/m2, QW
  Interventions: Drug: HCB101; Drug: Cetuximab; Drug: Pembrolizumab
- Cohort 6c: HCB101 + Cetuximab (Experimental): HCB101, QW Cetuximab 400 mg/m2 IV on D1, then 250 mg/m2, QW
  Interventions: Drug: HCB101; Drug: Cetuximab
- Cohort 7: HCB101 + Trastuzumab Deruxtecan (Experimental): HCB101, QW Trastuzumab Deruxtecan 5.4 mg/kg IV on D1, Q3W
  Interventions: Drug: HCB101; Drug: Trastuzumab deruxtecan
- Cohort 8: HCB101 + Atezolizumab/Toripalimab + Bevacizumab (Experimental): HCB101, QW Atezolizumab 1200 mg IV on D1, Q3W or Toripalimab 240 mg IV on D1, Q3W Bevacizumab 15 mg/kg IV on D1, Q3W
  Interventions: Drug: HCB101; Drug: Bevacizumab; Drug: Toripalimab; Drug: Atezolizumab
- Cohort 9: HCB101 + Atezolizumab/Toripalimab + carboplatin + etoposide. (Experimental): HCB101, QW Atezolizumab 1200 mg IV on D1, Q3W or Toripalimab 240 mg IV on D1, Q3W Carboplatin AUC=5, IV on D1, Q3W for 4 cycles Etoposide 100mg/m2, IV on D1, 2, 3, Q3W for 4 cycles
  Interventions: Drug: HCB101; Drug: Toripalimab; Drug: Carboplatin (AUC 5); Drug: Etoposide; Drug: Atezolizumab

INTERVENTIONS:
Drug: HCB101 — QW
Drug: Trastuzumab — 8 mg/kg IV loading dose on Day 1 of cycle 1, then 6 mg/kg IV every 21 days;
  Arms: Cohort 1: HCB101+Trastuzumab+Pertuzumab+CAPEOX
Drug: Pertuzumab — 840 mg IV on Day 1, cycled every 21 days;
  Arms: Cohort 1: HCB101+Trastuzumab+Pertuzumab+CAPEOX
Drug: Oxaliplatin — 130 mg/m2 IV on Day 1, cycled every 21 days
  Arms: Cohort 1: HCB101+Trastuzumab+Pertuzumab+CAPEOX; Cohort 3a: HCB101 + Bevacizumab + FOLFIRI/ mFOLFOX6; Cohort 3b: HCB101 + Cetuximab + FOLFIRI/ mFOLFOX6; Cohort 3d: HCB101 + mFOLFOX6; Cohort 5: HCB101 + Pembrolizumab + CAPEOX
Drug: Capecitabine — 1000 mg/m2 PO BID on Days 1-14, Cycled every 21 days
  Arms: Cohort 1: HCB101+Trastuzumab+Pertuzumab+CAPEOX; Cohort 5: HCB101 + Pembrolizumab + CAPEOX
Drug: Ramucirumab — 8 mg/kg IV on Days 1 and 15, Cycled every 28 days
  Arms: Cohort 2: HCB101+Ramucirumab+Paclitaxel; Cohort 3c: HCB101 + Ramucirumab + FOLFIRI
Drug: Paclitaxel — 80 mg/m2 IV on Days 1, 8, and 15, Cycled every 28 days
  Arms: Cohort 2: HCB101+Ramucirumab+Paclitaxel
Drug: Bevacizumab — 5 mg/kg IV on Day 1, Repeat every 2 weeks;
  Arms: Cohort 3a: HCB101 + Bevacizumab + FOLFIRI/ mFOLFOX6; Cohort 8: HCB101 + Atezolizumab/Toripalimab + Bevacizumab
Drug: Cetuximab — 400 mg/m2 first infusion, followed by 250 mg/m2 IV weekly;
  Arms: Cohort 3b: HCB101 + Cetuximab + FOLFIRI/ mFOLFOX6; Cohort 6b: HCB101 + Pembrolizumab + Cetuximab; Cohort 6c: HCB101 + Cetuximab
Drug: Irinotecan — 180 mg/m2 IV over 30-90 minutes on Day 1 every 2 weeks
  Arms: Cohort 3a: HCB101 + Bevacizumab + FOLFIRI/ mFOLFOX6; Cohort 3b: HCB101 + Cetuximab + FOLFIRI/ mFOLFOX6; Cohort 3c: HCB101 + Ramucirumab + FOLFIRI
Drug: Leucovorin — 400 mg/m2 IV on Day 1 every 2 weeks
  Arms: Cohort 3a: HCB101 + Bevacizumab + FOLFIRI/ mFOLFOX6; Cohort 3b: HCB101 + Cetuximab + FOLFIRI/ mFOLFOX6; Cohort 3c: HCB101 + Ramucirumab + FOLFIRI; Cohort 3d: HCB101 + mFOLFOX6
Drug: 5-FU — 400 mg/ m2 IV bolus on Day 1, followed by 1200 mg/m2/day x 2 days (total 2400 mg/m2 over 46-48 hours) IV continuous infusion Repeat every 2 weeks
  Arms: Cohort 3a: HCB101 + Bevacizumab + FOLFIRI/ mFOLFOX6; Cohort 3b: HCB101 + Cetuximab + FOLFIRI/ mFOLFOX6; Cohort 3c: HCB101 + Ramucirumab + FOLFIRI; Cohort 3d: HCB101 + mFOLFOX6
Drug: Toripalimab — 240 mg/kg IV on Day 1 Cycled every 21 days
  Arms: Cohort 4: HCB101 + Pembrolizumab/Toripalimab + albumin-bound paclitaxel; Cohort 8: HCB101 + Atezolizumab/Toripalimab + Bevacizumab; Cohort 9: HCB101 + Atezolizumab/Toripalimab + carboplatin + etoposide.
Drug: Albumin-bound paclitaxel — 125 mg/m2 IV on day 1 and Day 8 Cycled every 21 days
  Arms: Cohort 4: HCB101 + Pembrolizumab/Toripalimab + albumin-bound paclitaxel
Drug: Pembrolizumab — 200 mg IV day 1; given every 21 days
  Arms: Cohort 3a: HCB101 + Bevacizumab + FOLFIRI/ mFOLFOX6; Cohort 4: HCB101 + Pembrolizumab/Toripalimab + albumin-bound paclitaxel; Cohort 5: HCB101 + Pembrolizumab + CAPEOX; Cohort 6a: HCB101 + Pembrolizumab; Cohort 6b: HCB101 + Pembrolizumab + Cetuximab
Drug: Carboplatin (AUC 5) — AUC=5, IV on D1, Q3W for 4~6 cycles
  Arms: Cohort 9: HCB101 + Atezolizumab/Toripalimab + carboplatin + etoposide.
Drug: Etoposide — 100mg/m2, IV on D1, 2, 3, Q3W for 4~6 cycles
  Arms: Cohort 9: HCB101 + Atezolizumab/Toripalimab + carboplatin + etoposide.
Drug: Atezolizumab — 1200 mg IV on D1, Q3W
  Arms: Cohort 8: HCB101 + Atezolizumab/Toripalimab + Bevacizumab; Cohort 9: HCB101 + Atezolizumab/Toripalimab + carboplatin + etoposide.
Drug: Trastuzumab deruxtecan — 5.4 mg/kg IV on D1, Q3W
  Arms: Cohort 7: HCB101 + Trastuzumab Deruxtecan

SUMMARY:
This is a non-randomized, open-label, dose-escalation, and dose-expansion Phase Ib/IIa study to evaluate the safety, tolerability, PK, PD, and preliminary antitumor activity of HCB101 administered in combination with standard or approved anticancer therapies in subjects with advanced solid tumors. The trial includes a Part-I (Phase Ib) of the dose-escalation phase and a Part-II (Phase IIa) of the dose-expansion phase.

Part-I: Dose-escalation phase (Phase Ib):

Part I uses a standard 3+3 dose-escalation design to characterize safety and tolerability and to determine the maximum tolerated dose (MTD) and/or recommended Phase II dose (RP2D) of HCB101 when administered in combination regimens. The study includes 14 planned cohorts (Cohorts 1-9, including sub-cohorts 3a-3d and 6a-6c).

Part-II: Dose-expansion phase (Phase IIa) Based on safety, tolerability, PK/PD, and emerging antitumor activity observed in Part-I (Phase Ib), selected dose levels, tumor types, and combination regimens will be further investigated in Part-II (Phase IIa).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are able to understand and willing to provide signed informed consent.
2. Male and female subjects of ≥18 years of age, inclusive, at the time of signing the informed consent.
3. With histologically/cytologically confirmed diagnosis of advanced solid tumors as described below:

1) Cohort 1- Gastric Cancer, HER-Positive (First-Line): 2) Cohort 2 - Gastric Cancer (Second-Line): 3) Cohort 3 - Colorectal Cancer (Second-Line): 4) Cohort 4 - Triple-Negative Breast Cancer (First-Line): 5) Cohort 5 - Gastric Cancer, HER2 Medium/Low/Negative (First-Line): 6) Cohort 6 - Head and Neck Squamous Cell Carcinoma: 7) Cohort 7 - Ovarian Cancer: 8) Cohort 8 - Hepatocellular Carcinoma: 9) Cohort 9 - Extensive-Stage Small Cell Lung Cancer: 4. Have adequate organ function, as indicated by the following laboratory parameters below (had not received a blood transfusion, apheresis infusion, erythropoietin, granulocyte colony-stimulating factor, and other relevant medical support within 14 days before the administration of the first dose of study intervention).

Exclusion Criteria:

1. With a known history of hypersensitivity to any components of the study intervention.
2. Prior/Concomitant Therapy/Treatment:

   1. Subjects who have undergone major surgery or radical radiotherapy within 28 days before the first dose of study intervention.
   2. Subjects who have received systemic antitumor therapies within the following washout periods prior to the first dose of study intervention:

      * 28 days for curative radiotherapy, immunotherapy, or targeted therapy, etc.
      * 14 days for chemotherapy, palliative radiotherapy, endocrine therapy, or herbal medicine or traditional therapies with known or claimed antitumor activity.
   3. Subjects who have used a radioactive drug (Strontium, Samarium, etc.) within 56 days before the first dose of the study intervention.
   4. Subjects who are active using of vitamin K antagonist anticoagulant like warfarin. Use of low molecular weight heparin and factor Xa inhibitors will be permitted on a case-by-case basis. Daily low dose of aspirin use (≤ 100 mg QD in Mainland China; ≤ 81 mg QD in the United States) is allowed.
   5. Subjects who have received any treatment targeting the CD47 or SIRPα pathway.
   6. Subjects who have received or plan to receive live virus or bacterial vaccine within 28 days before the first dose of study intervention while the subject receives the study intervention.
3. Participation in another clinical study with an investigational product administered or investigational device used in the last 28 days (If half-life is not clear) or 5 half-lives (If half-life is clear, the longer time one prevails) before receiving the first dose of study intervention.
4. Subjects who have received any treatment targeting the CD47 or SIRPα pathway.
5. An uncontrolled acute infection.
6. Known to have a history of alcoholism or drug abuse.
7. Any other medical (e.g., Child-Pugh class B or C, pulmonary, metabolic, congenital, endocrinal or CNS disease, etc.), psychiatric, or social condition deemed by the Investigator to be likely to interfere with a subject's rights, safety, welfare or ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Number/incidence and percentage of subjects with adverse events. | 12 months
  To evaluate the safety and tolerability of HCB101
Number of subjects with Maximal tolerance dose (MTD) of HCB101 | 12 months
  To evaluate the tolerability of HCB101

SECONDARY OUTCOMES:
Overall Rate Response (ORR) | 12 months
  ORR is defined as the proportion of participants who have a partial response (PR) or critical response (CR)
Duration of Response (DoR) | 12 months
  DOR is defined as time from date of initial documentation of a response (PR or CR) to date of first documented evidence of progressive disease (PD)
Disease Control Rate (DCR) | 12 months
  DCR is defined as the proportion of participants who have a partial response (PR), critical response (CR), or disease stable (SD)
Progression-Free Survival (PFS) | 12 months
  Defined as the duration from the start of treatment until tumor progression or death of any cause.
Peak Plasma Concentration (Cmax) of HCB101 | 12 months
  Peak Plasma Concentration (Cmax) of HCB101 following single and repeated IV doses of HCB101 at different dose levels.
Area under the plasma concentration versus time curve (AUC) of HCB101 | 12 months
  Area under the plasma concentration versus time curve (AUC) of HCB101
Time to maximum drug concentration in plasma (Tmax) of HCB101 | 12 months
  Time to maximum drug concentration in plasma (Tmax) of HCB101 following single and repeated IV doses of HCB101 at different dose levels.
Terminal elimination half-life (t1/2) of HCB101 | 12 months
  Terminal elimination half-life (t1/2) of HCB101 following single and repeated IV doses of HCB101 at different dose levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No